CLINICAL TRIAL: NCT04625751
Title: Unravelling the Association Between Neurovascular Uncoupling and Autonomic Neuropathy in Patients With Type 2 Diabetes
Brief Title: Neurovascular Coupling and Autonomic Neuropathy in Type 2 Diabetes
Status: Active, not recruiting | Type: Observational
Sponsor: Hartwig R. Siebner (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Hartwig R. Siebner, Professor, DMSc, Danish Research Centre for Magnetic Resonance
Organization: Danish Research Centre for Magnetic Resonance (Other)
Other Study IDs: H-20031245
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes; Cardiovascular Autonomic Neuropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- T2DM +CAN
  Interventions: Other: CO2-enriched air; Other: Meal response test
- T2DM -CAN
  Interventions: Other: CO2-enriched air; Other: Meal response test
- Healthy control
  Interventions: Other: CO2-enriched air; Other: Meal response test

INTERVENTIONS:
Other: CO2-enriched air — To assess cardiovascular reactivity
Other: Meal response test — Meal response test to assess changes in splanchnic blood flow.

SUMMARY:
Diabetes is a growing global health care challenge. Diabetes patients may also suffer from cardiovascular autonomic neuropathy (CAN) which may affect cerebral perfusion. The main purpose of this project is to investigate the association between CAN and disturbances in the neurovascular coupling in type 2 diabetes patients. Moreover, the purpose is also to investigate coherence between CAN and the enteric nervous system. Finally, this project aims at delineating microstructural changes in the brain tissues as a consequence of CAN.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of type 2 diabetes (Patients)
* Age between 50-70 years (All)
* Presence of CAN as diagnosed by cardiovascular reflex tests with two or three pathological results (Patients with CAN only)
* Exclusion of CAN as diagnosed by cardiovascular reflex tests with no pathological results (Patients without CAN and HC only)

Exclusion Criteria:

* Participants receiving treatment with direct effects on noradrenergic or cholinergic signaling (for example beta-blockers, tricyclic antidepressants, SSRI's) (All)
* Acute infections (All)
* Thyroid disease (All)
* Substance or alcohol abuse (All)
* Atrial fibrillation or flutter (All)
* Respiratory failure (All)
* Participants in active laser treatment for retinopathy, will be excluded from the Valsalva test (Patients)
* Non-diabetic causes of neuropathy including a medical history of vitamin B12 deficiency, folic acid deficiency, rheumatoid arthritics, amyloidosis, HIV, syphilis, Borreliosis, drug induced neuropathy and neuropathy caused by toxins (All)
* Claustrophobia (All)
* Implanted pacemakers or remaining pacemaker electrodes (All)
* Previous heart or brain surgery with use of metal clips (All)
* Any form of non-MR-compatible implants
* Non-compliance with the study protocol as judged by the investigators (All)
* Concurrent participation in an intervention study (Patients)
* Participants who by judgments of the investigator, is incapable of participating (All)

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes and cardiovascular autonomic neuropathy. Patients with type 2 diabetes but no cardiovascular autonomic neuropathy Healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Neurovascular coupling | 1 hour
  Ratio between oxygen delivery/oxygen consumption by MRI during visual and hypercapnic stimulation
Cerebrovascular reactivity | 1 hour
  Change in CBF between normocapnia and hypercapnia
Structural differences in brain tissue | 1 hour
Regional splanchnic blood (superior mesenteric artery) flow increase in response to meal test | 3 hours
Change in blood levels of gastrointestinal hormones and markers of metabolism following meal test | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hartwig R. Siebner, MD, Prof, Principal Investigator — Danish Research Centre for Magnetic Resonance
Locations (2):
- Denmark (2):
  - Steno Diabetes Center Copenhagen, Gentofte Municipality
  - Danish Research Centre for Magnetic Resonance, Hvidovre

IPD SHARING:
Plan to Share IPD: Undecided